CLINICAL TRIAL: NCT06496139
Title: Emotion Regulation Based Internet-delivered Cognitive Behavioural Therapy for Premenstrual Dysphoric Disorder: A Randomised Controlled Trial
Brief Title: Emotion Regulation-based Internet-delivered Cognitive Behavioural Therapy for Premenstrual Dysphoric Disorder
Acronym: Premensis-s
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Utah State University (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-00655-01
Record Dates: First submitted 2024-05-29; First posted 2024-07-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Premenstrual Dysphoric Disorder
Keywords: Internet-delivered cognitive behavioural therapy; Emotion regulation; Premenstrual dysphoric disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The study is a parallel two-group randomised controlled trial with 1:1 allocation to 8 weeks of therapist-guided self-help ICBT (TG) or a waitlist control group (WL)
Who Masked: Outcomes Assessor
Masking Description: Randomisation will be performed externally by a person independent from the study. After group allocation, participants in the TG will be randomly assigned to one of the therapists involved in the trial. A statistician blinded to group allocation will conduct all statistical analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Therapist-guided self-help internet-delivered cognitive behavioural therapy for PMDD
  Interventions: Behavioral: Therapist-guided internet-delivered cognitive behavioural therapy
- Control group (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Therapist-guided internet-delivered cognitive behavioural therapy — The intervention consists of 8 weeks of therapist-guided self-help ICBT.
  Arms: Treatment group

SUMMARY:
Premenstrual dysphoric disorder (PMDD) is a debilitating cyclic mental disorder affecting about 2-5% of women of reproductive age. PMDD is characterised by recurring emotional, behavioural, cognitive, and somatic symptoms that arise during the luteal (premenstrual) phase of the menstrual cycle and remit shortly after the onset of menses. Although pharmacological interventions are available, many women experience residual symptoms, discontinue treatment or refrain from them because of side effects. Therefore, non-pharmacological treatment options are needed.

Preliminary evidence suggests that internet-delivered cognitive behavioural therapy (ICBT) is a promising candidate, but further research is warranted. Also, there is room for treatment improvement. Specifically, it has been suggested that components targeting emotional and interpersonal dysregulation should be incorporated into CBT for PMDD. The current study aims to assess the effects of an ICBT intervention for PMDD incorporating skills training in emotion regulation and interpersonal effectiveness in a randomised controlled trial (RCT).

DETAILED DESCRIPTION:
The study is a parallel two-group RCT with 1:1 allocation to 8 weeks of a therapist-guided self-help ICBT for PMDD or a waitlist control group. Approximately 164 women (age 18-45) fulfilling the DSM-5 diagnostic criteria for PMDD will be randomly assigned.

Recruitment

Participants will be recruited from the general population using the following screening procedure.

1. Web-based screening for PMDD (Premenstrual Screening Tool) and other eligibility criteria
2. Clinical diagnostic (telephone) interview assessing preliminary PMDD diagnosis and psychiatric comorbidity
3. Prospective daily ratings of premenstrual symptoms during two consecutive menstrual cycles using the Daily Report of Severity of Problems (DRSP).

Outcomes and Expected Results

Primary outcomes are pre- to post-treatment group differences in premenstrual symptoms and their impact on everyday life (prospective daily ratings, two menstrual cycles pre- and post-treatment) and PMDD-related psychological and functional impairment (retrospective ratings). Participants in the treatment group (vs waiting list) are expected to report a reduction in primary outcomes during the luteal (premenstrual) phase after treatment (vs baseline). No group differences in outcomes are expected during the follicular (post-menstrual) phase.

Secondary outcomes include treatment effects on quality of life (QoL) and difficulties in emotion regulation. Participants in the treatment group are expected to report higher QoL and lower levels of difficulties in emotion regulation after treatment (vs. baseline) than the waitlist control group. To assess long-term treatment effects, follow-up assessments will be conducted 6 and 12 months after treatment.

Health economic data will be collected for future health economic evaluations of the treatment.

Analysis

All randomised participants will be included in the intention-to-treat (ITT) population, regardless of whether they received or completed treatment. The per-protocol (PP) population will be a subgroup of the ITT population containing all participants without a major protocol violation. Sensitivity analyses will also be conducted with (1) participants who have completed at least four mandatory modules (modules 1-4) and (2) participants who have completed at least four mandatory modules and at least one of the optional lifestyle modules. To further explore potential differential effects of ICBT, exploratory analyses will be conducted for different symptom clusters (e.g., affective symptoms) and symptom trajectories in terms of onset and/or in combination with severity and severity peak. The relationship between difficulties in emotion regulation and improvement in primary outcomes will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. PMDD diagnosis according to DSM-5
2. Menstrual cycle length between 23-34 days, i.e., 5-8 cycles in the last six months
3. Sufficient proficiency in Swedish to comprehend the treatment materials
4. Access to computer/tablet/mobile phone with internet connection

Exclusion Criteria:

1. Breastfeeding or pregnancy during the previous three months
2. Initiation of or change in treatment with antidepressants, benzodiazepines, contraceptives, or hormones during the last three months
3. Current or history of a gynaecological disease (e.g., endometriosis, polycystic ovary syndrome) that may confound the results
4. Ongoing or previous psychological treatment for premenstrual disorders
5. Severe mental disorders that may interfere with the person's ability to complete the treatment or complicate the interpretation of results, e.g., psychosis, bipolar disorder, severe eating disorder, or severe depression
6. Elevated suicide risk (e.g., recurrent active suicidal ideation, current suicide plans, previous suicide attempts).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Group differences in premenstrual symptoms and their impact on everyday life during the luteal phase from baseline to post-treatment | Baseline to post-treatment (daily ratings over two menstrual cycles [ca 56 days] starting 8 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment (daily ratings one cycle [ca 28 days] beginning 6 and 12 months post-treatment).
  This primary outcome is assessed with the Daily Report of Severity of Problems. (DRSP) The DRSP assesses premenstrual symptoms included in DSM-5 diagnostic criteria for PMDD and their impact on everyday life. Items are rated on a scale from 1-6. Baseline and post-treatment data consist of prospective daily DRSP ratings over two consecutive menstrual cycles, both before and after treatment. Follow-up assessments will include daily DRSP ratings over one menstrual cycle.
Group differences in PMDD-related psychological and functional impairment during the luteal phase from baseline to post-treatment | Baseline to post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment. All assessements will be collected during luteal phase.
  This outcome is assessed using the PMS Impact Questionnaire (PMS-I) which includes two subscales: (1) psychological impairment and (2) functional impairment. The PMS-I consists of 18 items (9 for each subscale) rated on a scale from 1-4 scale (max score 72, higher points indicating higher levels of psychological and functional impairment).

SECONDARY OUTCOMES:
Group differences in quality of life during the luteal phase from baseline to post-treatment | Baseline to post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment. All assessements will be collected during luteal phase.
  Quality of life will be assessed using the Brunnsviken Brief Quality of Life scale (BBQ). The BBQ includes 12 items covering six life domains (recreation, philosophy of life, self-regard, creativity, learning and friendship), rated in terms of satisfaction and importance on scale from 0-4. Higher points indicate higher quality of life.
Group differences in difficulties in emotion regulation during the luteal phase from baseline to post-treatment. | Baseline to post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment. All assessements will be collected during luteal phase.
  Difficulties in emotion regulation will be assessed using the Difficulties in Emotion Regulation Scale (DERS-16). The DERS-16 measures five dimensions of emotion regulation in 16 items rated on a scale ranging from 1-5 (max score 80). High scores indicate more difficulties in emotion regulation.
Group differences in health-related quality of life during the luteal phase from baseline to post-treatment | Baseline to post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment. All assessements will be collected during luteal phase.
  Health-related quality of life will be assessed with the Assessing quality of life 8 dimensions (AQoL-8D). The AQoL-8D has 35 items and eight dimensions, including independent living, happiness, mental health, coping, relationships, self-worth, pain, and senses). Items have different response levels, each representing increasing levels of severity.
Remission (Full/Partial) | Post-treatment (daily ratings over two menstrual cycles [ca 56 days] starting 8 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment (daily ratings one cycle [ca 28 days] beginning 6 and 12 months post-treatment).
  Remission will be determined based on post-treatment DRSP symptom ratings over two menstrual cycles post-treatment using the C-PASS algorithm with a 30% change criterion. Full remission is defined as not fulfilling the criteria for PMDD or other menstrual-related mood disorders (MRMD) according to the C-PASS algorithm. Partial remission is defined as fulfilling the C-PASS algorithm for an MRMD but not for PMDD. Follow-ups: In the 6 and 12-month post-treatment follow-ups, remission will be based on the C-PASS algorithm applied to one menstrual cycle, as daily ratings will only be collected during one cycle at follow-ups.

OTHER OUTCOMES:
Treatment satisfaction (treatment group only) | Post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline)
  Satisfaction with treatment will be measured using the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 includes 8 items rated on a scale from 1-4 (max score 32, higher scores indicate higher satisfaction).
Treatment credibility and expectations (treatment group only) | Treatment week 2 and 4 (treatment is 8 weeks in total)
  The Credibility/Expectancy Questionnaire (CEQ) will be used to evaluate how treatment credibility and expectancy impact treatment effects. The CEQ includes 5 questions rated on a scale from 1-10 (max score 50; higher ratings indicate higher credibility and expectancy of positive treatment effects).
Negative effects of treatment (treatment group only) | Post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline)
  Negative effects of treatment will be assessed with the Negative Effects Questionnaire (NEQ). The NEQ includes 20 items rated on a scale from 0-4 (max 80, higher ratings indicating more negative effects)
Cost in relation to quality-adjusted life years (QALYs) | Baseline to post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment. All assessements will be collected during luteal phase.
  The QALY is a measure that comprises both quality of life and length of life and has an intrinsic value for money. QALYs will be estimated using individual scores from the Assessing quality of life 8 dimensions (AQoL-8D) and weights derived from the general population.
Societal resources used by participants | Baseline to post-treatment (first luteal phase after treatment, i.e., 8-10 weeks after baseline). Follow-up assessments at 6 and 12 months post-treatment. All assessements will be collected during luteal phase.
  The societal resources used by participants will be collected using an adapted version of the Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) questionnaire, assessed retrospectively for the past 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala university, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon reasonable request following trial completion and publication of results.
Supporting Information: Study Protocol, ICF, Analytic Code

REFERENCES:
- [Background] Reichwein JF, Patel MC, Pagenkopf BL. Rhodium-catalyzed regioselective olefin hydrophosphorylation. Org Lett. 2001 Dec 27;3(26):4303-6. doi: 10.1021/ol016989r. PMID 11784203
- [Derived] Hoppe JM, Weise C, Kleinstaeuber M, Skalkidou A, Vegelius J, Comasco E, Grondal M, Kaltsouni E, Sundstrom F, Sampaio F, Andersson G, Buhrman M. Emotion regulation-based internet-delivered cognitive behavioural therapy for premenstrual dysphoric disorder: study protocol for a randomised controlled trial in Sweden. BMJ Open. 2025 Jan 22;15(1):e091649. doi: 10.1136/bmjopen-2024-091649. PMID 39843366